CLINICAL TRIAL: NCT07352761
Title: Comparing Different Techniques of Bilateral Uterine Artery Occlusion During Laparoscopic Myomectomy: A Randomized Controlled Trial
Brief Title: Bilateral Uterine Artery Occlusion During Laparoscopic Myomectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Alexandria University, OBGYN
Record Dates: First submitted 2025-12-21; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-04

CONDITIONS: Uterine Fibroids (Leiomyoma); Myomectomy; Myomectomy; Surgical Blood Loss
Keywords: Fibroids; Laparoscopic myomectomy; Blood loss; Uterine artery occlusion; Ovarian reserve
MeSH Terms: conditions — Leiomyoma; Blood Loss, Surgical; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Temporary clipping of uterine arteries (Active Comparator)
  Interventions: Procedure: Temporary clipping of uterine artery
- Temporary occlusive suturing of uterine artery (Active Comparator)
  Interventions: Procedure: Temporary occlusive suturing of uterine artery
- Bipolar coagulation of uterine arteries (Active Comparator)
  Interventions: Procedure: Bipolar coagulation of uterine arteries
- No occlusion of uterine artery (Active Comparator)
  Interventions: Procedure: Laparoscopic myomectomy only

INTERVENTIONS:
Procedure: Temporary clipping of uterine artery — Both uterine arteries will be temporary clipped with a Titanium clip till the end of the myomectomy procedure
  Arms: Temporary clipping of uterine arteries
Procedure: Temporary occlusive suturing of uterine artery — A "Shoelace" suture will be applied to both uterine arteries and the sutures will be removed at the end of the myomectomy procdure
  Arms: Temporary occlusive suturing of uterine artery
Procedure: Bipolar coagulation of uterine arteries — Permanent coagulation of both uterine arteries will be performed by Bipolar forceps before the start of the myomectomy procedure
  Arms: Bipolar coagulation of uterine arteries
Procedure: Laparoscopic myomectomy only — No occlusion of uterine arteries will be performed. Only Laparoscopic myomectomy will be performed
  Arms: No occlusion of uterine artery

SUMMARY:
The current study is a multiple-arm, single blinded, and controlled randomized trial. It will be conducted in two gynecological endoscopy centers: • ElShatby University Hospital, a tertiary level hospital in Alexandria, Egypt. • Al-Madina Women Hospital, A specialized hospital of Obstetrics and Gynecology, Alexandria, Egypt. Patient selection: women with uterine leiomyomata and planning for laparoscopic myomectomy will be assessed for eligibility then will be enrolled in the trial according to the following inclusion and exclusion criteria, after providing a written informed consent of participation. Outcome variables of the study: The primary outcome is intraoperative blood loss and the change in postoperative hemoglobin. The secondary outcomes of this study are the operative time of performing uterine arteries occlusion and the postoperative ovarian reserve.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the safety and impact on ovarian reserve of different techniques of bilateral uterine artery occlusion in women in the reproductive age group scheduled for laparoscopic myomectomy. The main question[s] it aims to answer [is/are]:Do the different techniques for laparoscopic uterine artery occlusion prior to myomectomy decrease the intraoperative blood loss and the postoperative hemoglobin? The investigator intends to compare three different techniques for laparoscopic uterine artery occlusion (clipping, temporary suture, and coagulation) versus control group (no occlusion of uterine arteries) to see the effect on intraoperative blood loss, postoperative hemoglobin, and impact on ovarian reserve. Participants will be randomly allocated into one of the following study arms: * ARM 1: Will undergo temporary clipping of both uterine arteries before laparoscopic myomectomy (LAP-M). * ARM 2: Will undergo temporary occlusion of both uterine arteries using the Shoe-lace suture technique before LAP-M. * ARM 3: Will undergo permanent occlusion of both uterine arteries using bipolar coagulation before LAP-M. * ARM 4 (Control group): Will undergo only LAP-M without occlusion of uterine arteries.

ELIGIBILITY:
Inclusion Criteria:

* women with uterine fibroids and complaining of either abnormal uterine bleeding, infertility, urinary or rectosigmoid pressure manifestations.
* Fibroid size from 3 - 10 cm in diameter and with
* a maximum number of 3 fibroids.

Exclusion Criteria:

* contraindication to pneumoperitoneum and laparoscopy,
* patients with BMI > 30 kg/m2,
* history of midline abdominal incisions,
* women with history of prior ovarian surgery,
* women with history of hormonal treatment for the last 3 months before surgery,
* women who are not good candidate for myomectomy and who would benefit more from hysterectomy such as, women with multiple ≥ 4 leiomyomata, associated adenomyosis, recurrent fibroids after myomectomy.
* suspected endometrial malignancy or suspected leiomyosarcoma features on ultrasound and/or MRI.
* Submucous fibroids who will undergo hysteroscopic myomectomy beside the laparoscopic surgery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-identified females
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | Within 40 minutes of end of the myomectomy procedure
  The amount of intraoperative blood loss measured at the end of the procedure by estimation of the total volume of fluid in the suction machine.
Postoperative Hemoglobin shift | 24 hours after the procedure
  Postoperative hemoglobin level will be measured 24 hours after the procedure and the shift in hemoglobin from the preoperative level will be recorded

SECONDARY OUTCOMES:
Operative time of uterine artery occlusion | Time lapsed from intraperitoneal laparoscopic entry till completion of bilateral uterine artery occlusion (in minutes)
  Duration from accessing the retroperitoneum to occlusion of both uterine arteries
Total operative time | Time lapsed from intraperitoneal laparoscopic entry till completion of the myomectomy procedure and abdominal exit (in minutes)
  The total time lapse from the peritoneal entry till the end of the myomectomy procedure
Impact on ovarian reserve | 3 months postoperatively
  Serum AMH will be measured 3 months postoperative and compared with the preoperative level
Intraoperative complications | 40 minutes, 90 minutes, 120 minutes Intraoperative and 24 hours, 48 hours, 7 days Postoperatively
  The incidence of any intraoperative complications such as, blood transfusion, vascular injury, bowel injury, conversion to laparotomy, conversion to hysterectomy will be recorded in the four study arms.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Department of Obstetrics and Gynecology, Faculty of Medicine, Alexandria Univeristy, Alexandria, El-Shatby
  - • Al-Madina Women Hospital, A specialized hospital of Obstetrics and Gynecology, Alexandria, Egypt., Alexandria, Smouha

IPD SHARING:
Plan to Share IPD: No